CLINICAL TRIAL: NCT07306468
Title: Investigation of Exercise Capacity, Pulmonary Function, Respiratory Muscle Strength, and Quality of Life in Patients Diagnosed With Schizophrenia and Bipolar Disorder
Brief Title: Effects of Schizophrenia and Bipolar Disorder on Exercise Capacity, Pulmonary Function, and Quality of Life
Status: Recruiting | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Furkan Özdemir, Lecturer, Çankırı Karatekin University
Other Study IDs: 2025-06-26
Record Dates: First submitted 2025-11-25; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Schizophenia Disorder; Bipolar Disorder (BD)
Keywords: schizophrenia; bipolar disorder; respiratory functions; quality of life; exercise capacity
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Schizophrenia: Patients diagnosed with schizophrenia
  Interventions: Other: Pulmonary Function Test; Other: Respiratory Muscle Strength Evaluation; Other: Quality of Life Assessment; Other: Exercise Capacity Assessment
- Bipolar Disorder: Patients diagnosed with bipolar disorder
  Interventions: Other: Pulmonary Function Test; Other: Respiratory Muscle Strength Evaluation; Other: Quality of Life Assessment; Other: Exercise Capacity Assessment
- Healthy Control: Participants who have any diagnosed diseases/disorders
  Interventions: Other: Pulmonary Function Test; Other: Respiratory Muscle Strength Evaluation; Other: Quality of Life Assessment; Other: Exercise Capacity Assessment

INTERVENTIONS:
Other: Pulmonary Function Test — Participants' respiratory functions will assess with pulmonary function test according to ATS/ERS criteria
Other: Respiratory Muscle Strength Evaluation — Participants' respiratory muscle strenght will assess with maximal inspiratory pressure and maximal expiratory pressure assessment according to ATS/ERS criteria
Other: Quality of Life Assessment — Participants' quality of life will assess with WHOQOL-Bref questionnaire
Other: Exercise Capacity Assessment — Participants' exercise capacity will assess with 6 Minute Walk Test according to ATS/ERS criteria

SUMMARY:
This observational study aims to evaluate exercise capacity, pulmonary function, respiratory muscle strength, and quality of life in individuals diagnosed with schizophrenia and bipolar disorder. These psychiatric conditions are associated with sedentary lifestyles, metabolic side effects of psychotropic medications, and increased comorbidity risks, all of which may negatively impact physical fitness and respiratory health. By assessing cardiorespiratory endurance, pulmonary parameters (FVC, FEV₁), and respiratory muscle strength in this population, the study seeks to identify physiological limitations and contribute to the development of more effective rehabilitation strategies. The findings may support multidisciplinary approaches to improving physical health and overall quality of life in individuals with severe mental illness.

DETAILED DESCRIPTION:
Schizophrenia is a mental disorder observed in approximately 4 out of every 1,000 individuals in the general population, with a morbidity rate of 0.72%. According to the Global Burden of Disease Study (2010), around 20,000 deaths occur annually due to schizophrenia-related causes. Bipolar disorder is recognized as a chronic and severe mental illness. Based on data from the World Health Organization's global burden of disease reports, bipolar disorder ranks among the top 20 diseases contributing to disability worldwide and holds the 6th position among mental disorders.

Schizophrenia and bipolar disorder are serious and chronic psychiatric conditions affecting millions of individuals globally. The prevalence of schizophrenia is approximately 1%, while bipolar disorder has a lifetime prevalence of 2-3%. These disorders not only involve neuropsychiatric symptoms but also significantly impact physical health. In individuals with these conditions, sedentary lifestyle habits, metabolic side effects of antipsychotic and mood-stabilizing medications, and increased comorbidity risks are associated with notable reductions in exercise capacity.

Moreover, physical inactivity and heightened inflammatory processes may adversely affect respiratory muscle strength and pulmonary function. Studies have shown that patients with schizophrenia exhibit significantly lower maximal oxygen consumption (VO₂max) and anaerobic threshold levels compared to healthy individuals. In bipolar disorder, depressive episodes are marked by reduced exercise capacity, while manic episodes often involve irregular and risky physical activities.

Additionally, both disorders are associated with significantly lower pulmonary function parameters (FVC, FEV₁) compared to the healthy population. Respiratory muscle strength, a relatively underexplored area, is gaining importance. In schizophrenia cases dominated by negative symptoms, reduced inspiratory muscle strength combined with insufficient physical activity can severely limit patients' quality of life and independence. Similarly, in bipolar disorder, impairments in pulmonary capacity and respiratory muscle strength negatively affect quality of life.

Quality of life in these individuals is closely linked not only to mental health but also to physical capacity and pulmonary function. Enhancing respiratory muscle strength and aerobic capacity may positively influence overall quality of life, social participation, and functional status. However, the existing literature remains limited and fragmented. There is a noticeable lack of studies that simultaneously evaluate exercise capacity, pulmonary function, and respiratory muscle strength in individuals with psychiatric disorders.

This study aims to contribute to the literature from a multidisciplinary perspective by jointly examining exercise capacity, pulmonary function, respiratory muscle strength, and quality of life in individuals diagnosed with schizophrenia and bipolar disorder. These individuals often exhibit unhealthy lifestyle habits and a tendency toward sedentary behavior, which are considered risk factors that may adversely affect physical fitness. Components of physical fitness include cardiorespiratory endurance and muscular endurance. In light of this information, a review of the literature reveals that data on pulmonary function, respiratory muscle strength, and endurance in individuals with schizophrenia and bipolar disorder are still limited. The findings obtained from this study may guide the development of more effective rehabilitation and physical health support programs for these populations.

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer for participation
* Being 18 to 65 age

Exclusion Criteria:

* Having any respiratory, cardiac, neurologic or orthopedic disease which may affect respiratory functions or exercise capacity
* Having any neuropsychiatric disease except schizophrenia or bipolar disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals diagnosed with schizophrenia or bipolar disorder who are currently receiving standard medical treatment at the Community Mental Health Center of Çankırı State Hospital. Participants will be aged between 18 and 65 years, literate, and willing to participate in the study. No sampling method will be applied; all eligible individuals who meet the inclusion criteria and provide informed consent will be enrolled.
  Based on a prior sample size analysis conducted using data collected under approved ethical clearance, the study aims to include a total of 150 participants-50 individuals in each diagnostic group (schizophrenia, bipolar disorder and healthy controls). This sample size is expected to provide sufficient statistical power to detect differences between groups in terms of exercise capacity, pulmonary function, respiratory muscle strength, and quality of life.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Inspiratory Pressure (MIP) measurement | 1st day
  MIP will be measured using a mouth pressure device on Day 1 of the intervention. The maximum inspiratory pressure (MIP) will be recorded in cmH₂O. Three assessments will be performed, and the highest value will be reported.
Maximum Expiratory Pressure (MEP) measured in cmH₂O | 1st day
  MEP will be measured using a mouth pressure device on Day 1 of the intervention. The maximum expiratory pressure (MEP) will be recorded in cmH₂O. Three assessments will be performed, and the highest value will be reported.
Forced Expiratory Volume in 1 Second (FEV1) measured in liters | 1st day
  FEV1 will be measured using spirometry on Day 1 of the intervention. The maximum expiratory volume in 1 second (FEV1) will be recorded in liters. Three assessments will be performed, and the highest value will be reported.
Forced Vital Capacity (FVC) measured in liters | 1st day
  FVC will be measured using spirometry on Day 1 of the intervention. The forced vital capacity (FVC) will be recorded in liters. Three assessments will be performed, and the highest value will be reported.
FEV1/FVC ratio measured as a percentage | 1st day
  FEV1/FVC ratio will be calculated using spirometry on Day 1 of the intervention.
  The ratio of FEV1 to FVC will be expressed as a percentage. Three assessments will be performed, and the highest value will be reported.
Peak Expiratory Flow (PEF) measurement | 1st day
  PEF will be measured using spirometry on Day 1 of the intervention. The peak expiratory flow (PEF) will be recorded in liters per minute. Three assessments will be performed, and the highest value will be reported.

SECONDARY OUTCOMES:
6-minute walk distance (6MWD) measured in meters | 1st day
  The 6-minute walk test will be conducted according to standardized procedures in a straight corridor. Participants will be instructed to walk as far as possible in 6 minutes with standardized encouragement. The total distance walked will be recorded in meters. If a test is interrupted, the distance completed will be recorded. Two assessments will be performed on the same day, separated by a 30-minute rest interval. The 6-minute walk distance (6MWD) will be measured in meters, and the best (highest) distance will be reported.
WHOQOL-BREF total score measurement | 1st day
  Health-related quality of life will be assessed using the Turkish version of WHOQOL-BREF questionnaire. Participants will complete the 26-item survey at the 1st day. The total score will be calculated according to standardized scoring procedures and reported in points. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Çankırı, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No